CLINICAL TRIAL: NCT03032081
Title: High Intensity Interval Training in Heart Failure: The Gold Standard of Future Patient Care
Brief Title: High Intensity Interval Training in Heart Failure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI relocated, unable to complete the study. No replacement PI identified.
Sponsor: Georgia State University (Other)
Collaborators: Emory University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UL1TR000454 (NIH); CRN 00091835 (Other: Atlanta Clinical and Translational Science Institute)
Record Dates: First submitted 2017-01-24; First posted 2017-01-26 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Heart Failure; Physical Activity
MeSH Terms: conditions — Heart Failure; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Group (Experimental): 3 set of 4 minutes of cycling intense exercise, 4 days per week, for 8 weeks at about 80% to 90% of heart rate reserve
  Interventions: Other: High intensity exercise
- Moderate Intensity Group (Active Comparator): 40 to 47 minutes of continuous cycling exercise at 50% to 60% of heart rate reserve, 4 days per week, for 8 weeks.
  Interventions: Other: Moderate intensity exercise

INTERVENTIONS:
Other: High intensity exercise — High intensity exercise, defined as an exercise intensity of > 80% of heart rate reserve. Heart rate reserve is the maximum measured heart rate minus the measured resting heart rate.
  Arms: High Intensity Group
Other: Moderate intensity exercise — Moderate intensity exercise, defined as 50 to 60% of heart rate reserve for 40 to 47 minutes per day, 4 days per week, for 8 weeks. Heart rate reserve is the maximum measured heart rate minus the measured resting heart rate.
  Arms: Moderate Intensity Group

SUMMARY:
The investigators will assess the efficacy and safety of utilizing high-intensity interval training in stable heart failure patients on functional outcomes. Specifically, an assessment of baseline peak oxygen uptake and peak cardiac output will be assessed before and 8 weeks after intense interval training. Measurements of quality of life will be assessed before and after training as well as the number of arrhythmic events before and after training. The control group will be a group that will follow a moderate exercise training protocol over a similar period.

DETAILED DESCRIPTION:
Aerobic exercise training of moderate intensity is recommended as safe and effective for all stable outpatients with chronic heart failure who are able to participate in improving physical conditioning. Emerging data suggest that high-intensity exercise training in select heart failure patients may achieve even greater improvement in functional capacity than moderate intensity training leading to a better quality of life. In the few studies to date, aerobic capacity, heart function is increased to a better extent in heart failure patients that undergo an eight-week high-intensity exercise program (32 exercise sessions) compared to the standard of care. The goal of this pilot study is to collect data on safety and efficacy of high-intensity interval training in stable heart failure patients to demonstrate better physiological and clinical outcomes with fewer long-term health care costs compared to the standard of care. Twenty participants with stable heart failure (age range = 40 to 65 years of age) will be randomized into two different groups: the standard of care group, in which subjects will exercise for 40 minutes at 40 to 60 % of heart rate reserve (HRR) for eight weeks (32 sessions); and the high-intensity interval training group, in which subjects will perform four sets of 4-minutes at > 85% of HRR, with three minutes of active rest between intervals, for six weeks (32 sessions). The functional outcomes measured will be cardiac function (i.e. stroke volume, cardiac output, ejection fraction), pulmonary function (diffusing capacity, lung volumes, spirometry), exercise capacity (peak oxygen uptake) at rest and during exercise before and after eight weeks of exercise training (32 sessions). Adverse events related to each exercise training session (i.e. cardiac arrest, myocardial infarction during exercise, or within the first hour afterward) as well as arrhythmias will be recorded via Holter monitoring 24-hrs post-exercise. Quality of life will also be measured. The exercise training will be supervised at Grady Hospital. This novel approach has the chance to become impactful to these patients and will challenge the current negative perception of high-intensity exercise training in this patient population. The investigators anticipate this study will help reform the current exercise guidelines in these participants.

ELIGIBILITY:
Inclusion Criteria:

1. Stable, chronic heart failure with a left ventricular ejection fraction of 20 to 40%.
2. New York Heart Association (NYHA) class I to III symptoms with treatment that includes beta-blocker and angiotensin-converting enzyme (ACE) inhibitor and angiotensin receptor blocker (ARB) Therapy for at least eight weeks prior to exercise training if ejection fraction is < 35%.
3. No recent major cardiovascular hospitalizations or procedures within the previous three months.
4. Age 40-65 years
5. Aerobic capacity ≥ 12 mL/kg/min.
6. Subjects with an implantable cardioverter defibrillator (ICD) are also included.
7. Subjects with right ventricular systolic pressure ≤ 60 mmHg at rest.

Exclusion Criteria:

1. Inability to exercise (orthopedic or neurological problems).
2. History of seizure disorders.
3. History of atrial fibrillation or ventricular tachycardia in the past 3 months.
4. Implantable cardioverter defibrillator shocks due to atrial fibrillation or ventricular fibrillation within the past 3 months.
5. Presence of pacemaker.
6. Uncontrolled diabetes mellitus.
7. Diabetic insulin pump.
8. Uncontrolled hypertension.
9. Renal insufficiency (creatinine: > 2.5 mg/dl).
10. Severe left ventricular hypertrophy (> 1.8 cm wall thickness) or dynamic left ventricular outflow tract obstruction.
11. Greater than mild degree of valve stenosis or presence of an artificial heart valve.
12. Drug addiction.
13. Not being able to read and understand the consent form.
14. Signs of unreliableness.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2018-07-01 (Estimated); Study Completion 2018-07-01 (Estimated)

PRIMARY OUTCOMES:
Cardiac output | 8 weeks
  Measures how much blood is ejected from the left ventricle of the heart per minute (L/min). We will look at this at rest and at peak exercise.
Ejection fraction | 8 weeks
  Measures the fraction of blood ejected from the left ventricle at every heart beat (%). We will look at this at rest and at peak exercise.
Pulmonary diffusing capacity | 8 Weeks
  Measures gas transfer at the lung in mL/min/mmHg. We will look at this at rest and at peak exercise.

SECONDARY OUTCOMES:
Global longitudinal strain | 8 Weeks
  Measures measuring regional or global deformation of the heart measure in (number/s) at rest.
Heart rate variability | 8 weeks
  A measurement of either increased sympathetic or reduced vagal activity
Number of arrhythmic events | over a 24 hr period, before 8 weeks of training and after 8 weeks of training
  We are examining the number of times there is a recorded irregularity in the force or rhythm of the heartbeat.
Quality of Life | 8 weeks
  The MacNew Quality of Life questionnaire will be used to assess the emotional, physical, and social domains

CONTACTS AND LOCATIONS:
Overall Officials: Gerald S Zavorsky, PhD, Principal Investigator — Georgia State University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wisloff U, Stoylen A, Loennechen JP, Bruvold M, Rognmo O, Haram PM, Tjonna AE, Helgerud J, Slordahl SA, Lee SJ, Videm V, Bye A, Smith GL, Najjar SM, Ellingsen O, Skjaerpe T. Superior cardiovascular effect of aerobic interval training versus moderate continuous training in heart failure patients: a randomized study. Circulation. 2007 Jun 19;115(24):3086-94. doi: 10.1161/CIRCULATIONAHA.106.675041. Epub 2007 Jun 4. PMID 17548726
- [Background] Meyer P, Gayda M, Juneau M, Nigam A. High-intensity aerobic interval exercise in chronic heart failure. Curr Heart Fail Rep. 2013 Jun;10(2):130-8. doi: 10.1007/s11897-013-0130-3. PMID 23397179
- [Background] Flynn KE, Pina IL, Whellan DJ, Lin L, Blumenthal JA, Ellis SJ, Fine LJ, Howlett JG, Keteyian SJ, Kitzman DW, Kraus WE, Miller NH, Schulman KA, Spertus JA, O'Connor CM, Weinfurt KP; HF-ACTION Investigators. Effects of exercise training on health status in patients with chronic heart failure: HF-ACTION randomized controlled trial. JAMA. 2009 Apr 8;301(14):1451-9. doi: 10.1001/jama.2009.457. PMID 19351942
- [Background] Guiraud T, Labrunee M, Gaucher-Cazalis K, Despas F, Meyer P, Bosquet L, Gales C, Vaccaro A, Bousquet M, Galinier M, Senard JM, Pathak A. High-intensity interval exercise improves vagal tone and decreases arrhythmias in chronic heart failure. Med Sci Sports Exerc. 2013 Oct;45(10):1861-7. doi: 10.1249/MSS.0b013e3182967559. PMID 23591293
- [Background] Freyssin C, Verkindt C, Prieur F, Benaich P, Maunier S, Blanc P. Cardiac rehabilitation in chronic heart failure: effect of an 8-week, high-intensity interval training versus continuous training. Arch Phys Med Rehabil. 2012 Aug;93(8):1359-64. doi: 10.1016/j.apmr.2012.03.007. Epub 2012 Mar 21. PMID 22446291